An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

## 1.0 TITLE PAGE

**Drug Product** Desoximetasone 0.15% Topical Spray

**Design** An open label, safety study to assess the potential for adrenal

suppression following treatment with desoximetasone 0.15%

topical spray in patients with plaque psoriasis

**Population** Patients with a confirmed diagnosis of plaque psoriasis with 5-

10% body surface area affected

Patients will be enrolled in the following Cohorts:

• Cohort 1 - 12-18 years of age

• **Cohort 2** – 6-11 years of age

• Cohort 3 - 2-5 years of age

**Sponsor** Taro Pharmaceuticals U.S.A., Inc.

3 Skyline Drive

Hawthorne, NY 10532

Protocol Number DSXS 1503a

Novum Study Number 71615003

**IND** # 101789

Protocol Date 5/27/2016 Protocol Date Rev1 6/27/2016 Protocol Date Rev2 9/6/2016 NIIRB
September 13, 2016
APPROVED

This document is a confidential communication of Novum Pharmaceutical Research Services. Receipt of this document constitutes an agreement by the recipient that no unpublished information contained herein will be disclosed without Novum's written approval.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

## 2.0 KEY STUDY PERSONNEL AND FACILITIES

**Sponsor:** Taro Pharmaceuticals U.S.A., Inc.

3 Skyline Drive

Hawthorne, NY 10532

CRO: Novum Pharmaceutical Research Services (Novum)

225 W. Station Square Drive

Pittsburgh, PA 15219

**Sponsor's Representative:** Natalie Yantovskiy

Senior Director, Clinical Research Taro Pharmaceuticals U.S.A., Inc. 3 Skyline Drive, Hawthorne, NY 10532

Phone: 914-345-9001 Ext 6849

Fax: 914-593-0078

Email: Natalie.Yantovskiy@Taro.com

**CRO representative** Gail Gongas

Vice President, Clinical Trials

Novum Pharmaceutical Research Services

Tel: 412-363-3300 x 522 Fax: 412-924-0522

Email: gdgongas@novumprs.com

Medical Monitor: Paolo Fanzio, MD

Medical Monitor

Novum Pharmaceutical Research Services

Tel: 412-363-3300 x 597 Fax: 412-291-3171

Email: pmfanzio@novumprs.com

Biostatistician: Jianhua Liu, MSc

Senior Biostatistician

Novum Pharmaceutical Research Services

Tel: 647-779-6883

Email: jliu@novumprs.com

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# SIGNATURE PAGE

We, the undersigned, have carefully read this protocol and agree that it contains all the necessary information required to conduct the study. The study will be performed according to this protocol, all applicable FDA regulations, ICH guidelines and Good Clinical Practice standards.

| Gail Gongas Vice President, Clinical Trials Novum Pharmaceutical Research Services | 09/16/16<br>Date |
|---|---|
| Paolo Fanzio, MD Medical Monitor Novum Pharmaceutical Research Services | 9/23/2016<br>Date |
| Keith D. Gallicano, PhD Vice President, Scientific Affairs Novum Pharmaceutical Research Services | 09/19/2016<br>Date |
| N. Yantovskiy Natalie Yantovskiy | 27 Sep 2016 Date |

Senior Director, Clinical Research Taro Pharmaceutical USA, Inc.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# PRINCIPAL INVESTIGATOR'S SIGNATURE

| Iaccordance with FDA regulations, ICH deviations from the protocol may be Pharmaceuticals, USA) or Novum Pharma | guidelines and Good C<br>made without the price | or permission of the | derstand that no<br>Sponsor (Taro |
|---|---|---|---|
| Principal Investigator | _ | Date | |

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# 3.0 TABLE OF CONTENTS

| 1.0 | TITL | E PAGE | 1 |
|------|-------|-------------------------------------------------------|----|
| 2.0 | KEY | STUDY PERSONNEL AND FACILITIES | 2 |
| SIGN | ATURI | E PAGE | 3 |
| 3.0 | TABI | LE OF CONTENTS | 5 |
| 4.0 | SYNO | OPSIS | 8 |
| 5.0 | STUI | DY SCHEMATIC | 13 |
| 6.0 | LIST | OF ABBREVIATIONS AND TERMS | 14 |
| 7.0 | INTR | ODUCTION | 15 |
| 7.1 | Dis | sease Being Treated | 15 |
| 7.2 | Av | ailability and Efficacy of Already Approved Therapies | 16 |
| 7.3 | Sci | entific and Statistical Considerations | 16 |
| 7.4 | Ris | sks and Benefits | 17 |
| 8.0 | STUI | DY OBJECTIVES | 17 |
| 9.0 | INVE | ESTIGATIONAL PLAN | 17 |
| 9.1 | Stu | ndy Design and Plan Description | 17 |
| 9.2 | Sel | lection of Study Design | 18 |
| 9.3 | Sel | lection of Study Population | 19 |
| 9 | .3.1 | Inclusion Criteria | 19 |
| 9 | .3.2 | Exclusion Criteria | 19 |
| 9 | .3.3 | Restrictions during the Study | 20 |
| 9 | .3.4 | Removal of Patients from the Study | 21 |
| 9.4 | Tre | eatments | 22 |
| 9 | .4.1 | Treatments Administration | 22 |
| 9 | .4.2 | Identity of Investigational Product | 23 |
| 9 | .4.3 | Method of Assigning Patients to Treatment Groups | 23 |
| 9 | .4.4 | Packaging | 23 |
| 9 | .4.5 | Accountability | 23 |
| 9 | .4.6 | Compliance | 24 |
| 9.5 | Stu | ldy Conduct | 24 |
| 9 | .5.1 | Visit 1 (Day 1): Screening/Enrollment, Before 12 pm | 24 |

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

| 9.5.2 | Visit 2 (Day 14 ± 2): Interim Visit | 25 |
|---|---|---|
| 9.5.3 | Visit 3 (Day 29 ± 2): End of Study or Early Termination, Before 12 pm | 26 |
| 9.5.4 Vi | isit 4 (Day 42 ± 4): Follow-up Phone Call | 26 |
| 9.6 Stu | idy Procedures | 26 |
| 9.6.1 | Informed Consent | 26 |
| 9.6.2 | Demographics | 27 |
| 9.6.3 | Medical History | 27 |
| 9.6.4 | Vital Signs | 27 |
| 9.6.5 | Physical Exam and % Body Surface Area (BSA) | 27 |
| 9.6.6 | Application Site Reaction Assessment | 27 |
| At Visit | s 1, 2 and 3, the application site reactions will be recorded (see Appendix C) | 27 |
| 9.6.7 | Investigator Global Assessment | 27 |
| 9.6.8 | Concomitant Medication Use | 27 |
| 9.6.9 | Pregnancy Test | 27 |
| 9.6.10 | Dispensing Study Drug | 28 |
| 9.6.11 | Collecting Study Drug | 28 |
| 9.6.12 | Dosing Instructions and Diary | 28 |
| 9.6.13 | Dosing Compliance | 28 |
| 9.6.14 | Standard Sunscreen and Patient Wristband | 28 |
| 9.6.15 | Laboratory Evaluation | 28 |
| 9.6.16 | Cortisol Response Test. | 28 |
| 9.7 Ad | verse Events | 30 |
| 9.7.1 | Adverse Event Definitions | 30 |
| 9.7.2 | Severity of Adverse Event | 30 |
| 9.7.3 | Relationship of Adverse Event | 30 |
| 9.7.4 | Patient Participation Stopping Criteria | 31 |
| 9.8 Ser | rious Adverse Events | 31 |
| 9.8.1 | Definition of a Serious Adverse Event | 31 |
| 9.8.2 | Reporting Serious Adverse Events | 31 |
| 10.0 STA | FISTICAL METHODS | 32 |
| 10.1 Sta | itistical Plan | 32 |
| 10.1.1 | Determination of Sample Size | 32 |

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

| 10.1.2 Baseline Comparability | 33 |
|-----------------------------------------------------------|----------------|
| 10.1.3 Safety Analysis of Potential HPA Axis Suppression | 33 |
| 10.2 Safety Analysis | 33 |
| 11.0 REGULATORY OBLIGATIONS | 34 |
| 11.1 Institutional Review Board | 34 |
| 11.2 Study Documentation | 34 |
| 11.2.1 Protocol | 34 |
| 11.2.2 Informed Consent | 34 |
| 11.2.3 Protocol and Informed Consent Changes | 35 |
| 11.2.4 Source Documents and Case Report Forms | 35 |
| 11.2.5 Drug Accountability | 35 |
| 11.2.6 Drug Storage | 35 |
| 11.2.7 Pregnancies | 35 |
| 11.2.8 Reporting Safety Information to the IRB | 36 |
| 11.2.9 Record Retention. | 36 |
| 11.2.10 Study Monitoring and Auditing | 36 |
| 11.2.11 End of the Trial | 36 |
| 11.2.12 Clinical Study Report | 37 |
| 12.0 REFERENCES | 38 |
| 13.0 APPENDICES | 39 |
| APPENDIX A: Body Surface Area Calculation | 39 |
| APPENDIX B: Investigator Global Assessment (IGA) | 41 |
| APPENDIX C: Application Site Reactions | 42 |
| APPENDIX D: Cortisol Response Test | 43 |
| APPENDIX E: Evaluation of HPA Axis Suppression | 45 |
| APPENDIX F: Clinical Laboratory Testing | 46 |
| APPENDIX G: Cortrosyn <sup>TM</sup> Package Insert | 47 |
| APPENDIX H: Investigator Brochure, Desoximetasone 0.15% T | opical Spray50 |
| APPENDIX I: Protocol Revisions | 51 |

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# 4.0 SYNOPSIS

| Protocol Number | DSXS 1503a |
|---|---|
| Title | An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis |
| Objectives | <ol> <li>The objective of this study is to evaluate the potential of desoximetasone 0.15% topical spray to suppress HPA axis function in patients with mild to moderate plaque psoriasis.</li> <li>The secondary objectives are to evaluate the efficacy parameters and adverse event (AE) profile of desoximetasone 0.15% topical spray administered to patients with mild to moderate plaque psoriasis.</li> </ol> |
| Sponsor | Taro Pharmaceuticals U.S.A., Inc. |
| Name of Test<br>Product | Desoximetasone 0.15% Topical Spray |
| Route of<br>Administration | Topical |
| Study Design | An open label, safety study to assess the potential for adrenal suppression following treatment with desoximetasone 0.15% topical spray administered twice daily for 28 days in patients with mild to moderate plaque psoriasis. |
| Study Population | Approximately twenty five (25) to fifty (50) patients, stratified by age with a confirmed diagnosis of mild to moderate plaque psoriasis with: Cohort 1 – 10-20 patients age 12-18 years of age with 5-10% BSA affected Cohort 2 – 10-20 patients age 6-11 years of age with 5-10% BSA affected Cohort 3 – 5-10 patients age 2-5 years of age with 5-10% BSA affected Cohorts will be enrolled in sequential order. Each cohort will initiate enrollment once the previous cohort has reached the minimum number of patients and a safety analysis has been reviewed. Each cohort will be enrolled based on the availability of patients. |
| | Each cohort will be reviewed for the potential of HPA axis suppression. If at least 50% of patients in a cohort experience HPA axis suppression once the minimum number of patients has been enrolled and completed the cohort, enrollment for that cohort will be stopped and no further cohorts will be initiated. If at least 35% of patients have experienced HPA axis suppression across cohorts combined during the study, enrollment will be discontinued |

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

| Study Conduct | and no other cohorts will be initiated. Cohort 2 will not begin until safety data has been reviewed for Cohort 1. The same process will be followed for each Cohort until the study is complete. The enrollment in the individual Cohort may not be required if the satisfactory safety data for the same age group was obtained in the study DSXS 1503. All patients will attend the clinic for 3 scheduled visits: Visit 1: Screening/Enrollment (Day 1) Visit 2: Interim Visit (Day 14 ± 2) |
|---|---|
| | <b>Visit 3:</b> End of Study (Day $29 \pm 2$ ) or Early Termination |
| Inclusion Criteria | 1. Male or non pregnant, non lactating females: |
| | <ul> <li>Cohort 1 – 12-18 years of age</li> <li>Cohort 2 – 6-11 years of age</li> <li>Cohort 3 – 2-5 years of age</li> </ul> |
| | 2. If female and of child bearing potential, have a negative urine pregnancy test at the baseline/ randomization visits and prepared to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g., condom with spermicide, IUD, oral, injected, transdermal or implanted hormonal contraceptives). |
| | 3. Signed informed consent form which meets all current ICH/FDA regulations. For patients under the age of majority in the state the study is being conducted (18 years in most states) the parent or legal guardian should sign the consent form and the child will be required to sign a patient "assent" form that will be written in such a way as to be understandable to a child. |
| | Based on the patient's age 11 -17 years old will read and sign an IRB approved assent form. Patients 6-10 years of age will provide verbal assent to participate. |
| | 4. Patients with a definite clinical diagnosis of stable plaque psoriasis: |
| | <ul> <li>Cohort 1 –age 12-18 years of age with 5-10% BSA affected (excluding face and scalp)</li> <li>Cohort 2 –age 6-11 years of age with 5-10% BSA affected (excluding face and scalp)</li> <li>Cohort 3 –age 2-5 years of age with 5-10% BSA affected (excluding face and scalp)</li> </ul> |
| | 5. Investigator Global Assessment (IGA) score of 2 (mild) or 3 (moderate) at baseline (see Appendix B) for the overall disease severity. |

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

## **Exclusion Criteria**

- 1. Patients under 2 years of age.
- 2. Females who are pregnant, lactating or likely to become pregnant during the study, or if of child-bearing potential and sexually active not willing to use appropriate contraceptive methods to avoid pregnancy.
- 3. Plaque psoriasis with a BSA involvement of < 5% or > 10%.
- 4. Investigator Global Assessment (IGA) of less than 2 (mild) or greater than 3 (moderate) at baseline.
- 5. Current diagnosis of types of psoriasis other than stable plaque psoriasis (i.e., erythrodermic, exfolative or pustular psoriasis).
- 6. Patient who will require active treatment with a restricted medication during the study.
- 7. History of psoriasis that has been unresponsive to topical corticosteroid therapy.
- 8. In the Investigator's opinion, the patient has other dermatological conditions, such as atopic or contact dermatitis, that may interfere with the clinical assessments of the signs and symptoms of psoriasis.
- 9. History of allergy or sensitivity to corticosteroids or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the patient or the results of the study.
- 10. History of an adverse reaction to Cortrosyn<sup>TM</sup> or similar test reagents.
- 11. Significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participation in the study.
- 12. Any radiation therapy, anti-neoplastic agents or immunosuppressant medication within 4 weeks before the first dose of study drug.
- 13. Treatment with any systemic antipsoriatic therapy or phototherapy (UVB or UVA) within 8 weeks before the first dose of study drug.
- 14. Treatment with any biological therapies for psoriasis within 12 weeks (or five half-lives whichever is less) before the first dose of study drug.
- 15. Treatment with any systemic steroids within 4 weeks of the first dose of the study drug. The use of inhaled or intranasal corticosteroids is acceptable as long as usage has been stable for at least 2 weeks before the first dose of study drug and will be continued during the

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

| | study. |
|---|---|
| | 16. Use of any topical antipsoriatic agents of any kind or any topical corticosteroids for any reason within 2 weeks before first use of study drug. Nonprescription antipsoriatic shampoos used only on the scalp will be allowed during the study. |
| | 17. Inability to understand the protocol requirements, instructions, and study-related restrictions, the nature, scope, and possible consequences of the clinical study. |
| | 18. Unlikely to comply with the protocol requirements, instructions, and study-related restrictions, such as uncooperative attitude, inability to return for follow-up visits, and improbability of completing the clinical study. |
| | 19. Receipt of any drug as part of a research study within 30 days before first dosing. |
| | 20. The patient is a member of the investigational study staff or a member of the family of the investigational study staff. |
| | 21. Previous participation in this study including patients previously enrolled in DSXS 1503. |
| Criteria for<br>Evaluation | Primary Outcome Measures: Hypothalamic Pituitary Adrenal (HPA) Axis Response to Cosyntropin demonstrating the absence or presence of adrenal suppression at the end of |
| | treatment Secondary Outcome Measures: Hypothalamic Pituitary Adrenal (HPA) Axis Response to Cosyntropin demonstrating the presence of adrenal suppression at the end of treatment with %BSA as a covariate |
| HPA Axis<br>Evaluation | Prior to the first dose of study drug and at the end of the study (Day 28 or early termination) all patients will have a cortisol response test performed using the procedure of Wood et al. (See Appendix D). Only those patients with normal adrenal function at baseline will be enrolled and dispensed study drug. If at the end of the study the patient has a cortisol response test that is suggestive of HPA axis suppression, they will have an additional test at least every 4 weeks until such time as the Investigator considers the adrenal function has returned to normal. |
| | Cohorts will be enrolled in sequential order. Each cohort will initiate enrollment once the previous cohort has reached the minimum number of patients and a safety analysis has been reviewed. Each cohort will be enrolled based on the availability of patients. |
| | Each cohort will be reviewed for the potential of HPA axis suppression. If at |

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

| | least 50% of patients in each Cohort experience HPA axis suppression once the minimum number of patients has been enrolled and completed the cohort, enrollment for that cohort will be stopped and no further cohorts will be initiated. If at least 35% of patients have experienced HPA axis suppression across cohorts combined during the study, enrollment will be discontinued and no other cohorts will be initiated. Cohort 2 will not begin until safety data has been reviewed for Cohort 1. The same process will be followed for each Cohort until the study is complete. |
|---|---|
| | Primary Analysis: Proportion of patients in the study with HPA axis suppression following treatment with the study medication. |
| | Secondary Analysis: |
| | A logistic regression of the proportion of patients in the study with HPA axis suppression will be performed with % BSA affected as a covariate. |
| Safety Parameters | Adverse events will be classified using standard MedDRA terminology Version 19.0 or higher and summarized by treatment group. Summary tables comparing the type, incidence, severity and Investigator's opinion of relationship to the study drug will be prepared by treatment group. Signs and symptoms of psoriasis will not be considered adverse events, unless in the Investigator's opinion, they have increased in frequency and/or severity to such an extent that the Investigator/patient considers that it is in the patient's best interest to be dropped from continued participation in the study and given alternative therapy for their condition. |
| | If sufficient data exist, adverse event frequencies will be compared between treatments using Fisher's exact test or a similar test. Concomitant medication use during the study will be tabulated by patient. |
| | Adverse events reported during the study will be tabulated in a summary table listing the type, incidence, severity and Investigator's opinion to drug relationship. |
| Sample Size<br>Determination | The sample size of 25 to 50 patients, stratified by age and % BSA, was determined to be sufficient for the study. |

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# 5.0 STUDY SCHEMATIC

| | Visit 1 | Visit 2 | Visit 3 | Visit 4 |
|---|---|---|---|---|
| Day | 1 | 14 ± 2 | 29 ± 2 | 42 ± 4 |
| Procedures | Screening/<br>Enrollment<br>Before 12 pm | Interim<br>Visit | End of Study/Early Termination Before 12 pm | Telephone<br>Follow-Up<br>Visit |
| Informed Consent | X | | | |
| Medical History and<br>Demographics | X | | | |
| Vital Signs | X | X | X | |
| Pregnancy Test* | X | X | X | |
| Physical Exam | X | | X | |
| % BSA Assessment | X | X | X | |
| IGA Score | X | X | X | |
| Application Site Reaction<br>Assessment | X | X | X | |
| Concomitant Medication | X | X | X | |
| Laboratory Evaluations | X | | X | |
| Cortisol Response Test | X | | X | |
| Confirm<br>Inclusion/Exclusion<br>Criteria | X | | | |
| Dispense Sunscreen and<br>Wristband | X | | | |
| Weigh and Dispense Study<br>Drug | X | X | | |
| Collect and Weigh Study<br>Drug | | X | X | |
| Dispense/Review Patient<br>Diary | X | X | X | |
| Adverse Events | | X | X | X |
| Evaluation of Patient<br>Compliance to the Protocol | | X | X | |

<sup>\*</sup> Pregnancy test will be carried out for females of childbearing potential.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# 6.0 LIST OF ABBREVIATIONS AND TERMS

| Abbreviation | Term |
|--------------|-------------------------------------------|
| ADL | Activities for Daily Living |
| ADR | Adverse Drug Reaction |
| AE | Adverse Event |
| BP | Blood Pressure |
| С | Celsius |
| CRF | Case Report Form |
| CRO | Clinical Research Organization |
| eCTD | electronic Common Technical Document |
| FDA | Food and Drug Administration |
| HR | Heart Rate |
| HRT | Hormone Replacement Therapy |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| IGA | Investigator's Global Assessment |
| IND | Investigational New Drug |
| IRB | Institutional Review Board |
| ITT | Intent-to-Treat |
| IUD | Intrauterine Device |
| LOCF | Last Observation Carried Forward |
| ml | Milliliter |
| mITT | Modified Intent-to-Treat |
| NDA | New Drug Application |
| NSAID | Non-Steroidal Anti-Inflammatory Drug |
| OHRP | Office of Human Rights Protection |
| OTC | Over-the-Counter |
| PUVA | Psoralen and UltraViolet A |
| RR | Respiratory Rate |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| USA | United States of America |

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

## 7.0 INTRODUCTION

Taro Pharmaceuticals U.S.A., Inc. (Taro) plans to submit an Investigational New Drug Application (IND) for a new formulation of desoximetasone; desoximetasone 0.15% topical spray. This product contains a potent corticosteroid to be indicated for the treatment of plaque psoriasis in patients 2 years of age or older.

# 7.1 Disease Being Treated

Psoriasis is an immune (T-cell)-mediated inflammatory skin disease that affects approximately 2% of the western population.<sup>1</sup> The most common type of psoriasis in both adults and children is plaque psoriasis, which is characterized by the presence of raised, thickened red lesions that are covered by silvery white scales, most commonly seen on the knees and/or elbows. Although there are reports implicating a genetic association with the disease, there are also studies that have established a set of psoriasis triggers including stress, medications (such as lithium, antimalarials, indomethacin, quinidine, beta blockers), injury or infection. The condition is considered chronic although the frequency and severity of outbreak in an individual can fluctuate without apparent cause.<sup>1-3</sup>

Treatment of plaque psoriasis depends on the severity of the condition, previous treatment regimens and personal preference of the patient. For mild to moderate plaque psoriasis, topical treatments and phototherapy are the preferred treatment modalities. For more severe cases oral or injectable systemic therapy may be warranted; however, the side effect profile of these products limits their use.

In some instances high potency steroids applied topically have been known to cause suppression of the hypothalamic-pituitary-adrenal (HPA) axis. In order to assess HPA axis function plasma levels of cortisol are measured prior (basal) and after a bolus administration of synthetic α 1-24-adrenocorticotropic hormone (ACTH). In this study Cortrosyn<sup>TM</sup> (cosyntropin, a synthetic subunit of ACTH) (Amphstar Pharmaceuticals, Inc.) will be used according to manufacturer instructions to assess HPA axis function (See Appendices D, E).<sup>4</sup> Recovery from steroid-induced adrenal insufficiency is usually rapid after the treatment is withdrawn.<sup>5</sup> See Appendix E for further explanation of the evaluation of the role of topical corticosteroids in HPA axis suppression.

Taro Pharmaceuticals USA has recently completed an open label safety and efficacy study to assess adrenal suppression in adults with moderate to severe plaque psoriasis after 4 weeks of treatment under maximal use conditions with the test product, desoximetasone 0.25% spray. Of 21 evaluable subjects, adrenal suppression was identified in 1 of 12 subjects having involvement of 10-15% of body surface area (BSA) and 2 of 9 subjects having involvement of > 15% of BSA after treatment with Topicort® Topical Spray twice a day for 28 days. Adrenal function returned to normal at the first follow-up visit, which was 28 days after the end of treatment, for all 3 of these patients<sup>6</sup>

This study design is based on similar studies performed, submitted and accepted by the FDA for recently approved high potency spray and foam topical corticosteroid formulations, topical corticosteroid/topical vitamin D3 analogue combination agents, and based on recommendations

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

provided by the FDA in IND 101789 Guidance Meeting (01/14/2015, Reference ID 3689041), regarding the scope and design of studies for desoximetasone 0.15% spray and an FDA Advice Letter dated 04/27/2015. 4,7,8,9,10,14

# 7.2 Availability and Efficacy of Already Approved Therapies

Treatment of plaque psoriasis depends on the severity of the condition, previous treatment regimens and personal preference of the patient. Psoriasis treatments historically include topical creams, sprays, lotions, foams or the more recently introduced-shampoos. Examples of marketed products include corticosteroids (Topicort<sup>®</sup>, Clobex<sup>™</sup>), Vitamin A & D derivatives (Tzorac<sup>®</sup>, Dovonex<sup>®</sup>), NSAIDs (salicylic acid), etc. For more severe cases, systemic therapy (methotrexate, oral retinoids, UV light, biologics etc) may be warranted; however, the side effect profile of these products limits their use.<sup>1,2,4,11,12</sup>

Desoximetasone is a high potency synthetic corticosteroid marketed in a number of formulations: gel (0.05%), cream (0.05% and 0.25%), and ointment (0.05% and 0.25%). All these formulations are encompassed under the Topicort® brand, acquired by Taro Pharmaceuticals U.S.A., Inc. (Taro) in 2004. Most recently, Taro received approval on April 11, 2013 for a new dosage form (spray) under NDA #204141, Topicort® (desoximetasone) Topical Spray, 0.25%, a super high potency formulation that is indicated for the treatment of plaque psoriasis in patients 18 years of age or older.

A new formulation of desoximetasone - Desoximetasone 0.15% Topical Spray has been developed by Taro Pharmaceuticals U.S.A., Inc. (Taro), and is the Test product used in this study.

## 7.3 Scientific and Statistical Considerations

Taro Pharmaceuticals USA, Inc. has developed and marketed Topicort <sup>®</sup> (desoximetasone 0.25%) topical spray, and Topicort <sup>®</sup> (desoximetasone 0.25% & 0.05%) topical creams, for the treatment of plaque psoriasis. <sup>11</sup> Topical application of high potency steroids at the recommended dosing levels are usually well tolerated in all populations, with less than 2% of patients reporting adverse reactions (7% in the pediatric population). The most commonly reported adverse events are burning, stinging, pruritus, and skin thinning/atrophy. <sup>1,2,4,11,12</sup>

In some instances high potency steroids applied topically have been known to cause suppression of the hypothalamic-pituitary-adrenal (HPA) axis. In order to assess HPA axis function plasma levels of cortisol are measured before (basal) and after a bolus administration of synthetic  $\alpha$  1-24-adrenocorticotropic hormone (ACTH). In this study Cortrosyn<sup>TM</sup> (cosyntropin, a synthetic subunit of ACTH) (Amphstar Pharmaceuticals, Inc.) will be used according to manufacturer instructions to assess HPA axis function (See Appendices D, E).<sup>4</sup> Recovery from steroid-induced adrenal insufficiency is usually rapid after the treatment is withdrawn.<sup>5</sup> See Appendix E for further explanation of the evaluation of the role of topical corticosteroids in HPA axis suppression.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

#### 7.4 Risks and Benefits

Known adverse reactions to topical corticosteroids include burning, itching, irritation, dryness, folliculitis, hypertrichosis, acneiform eruptions, hypopigmentation, perioral dermatitis, allergic contact dermatitis, maceration of the skin, secondary infection, skin atrophy, striae and milliaria. Dosing for extended periods of time may result in suppression of adrenal function.

Cortrosyn<sup>TM</sup> for injection is intended diagnostic and not therapeutic use and adverse reactions other than a rare hypersensitivity reaction are not anticipated. Known reactions are slight whealing with erythema at the site of injection.

The subject may benefit from clearing of the lesions and improvement of the condition of the disease. If the drug is approved, then many children may benefit from its use.

The potential risks and benefits of participation in the study will be explained to the patient and parent or legal guardian verbally and written in the informed consent form.

All patients enrolled in this study will receive the benefit of free specialized medical care, beyond standard medical treatment that would be expected through most health insurance plans. In addition, the patient will receive a stipend as compensation for time and inconvenience related to study participation including costs associated with travel to and from the medical facility.

Ethical consideration related to this protocol and the use of human patients will be reviewed by an IRB.

## 8.0 STUDY OBJECTIVES

- 1. The primary objective of this study is to evaluate the potential of desoximetasone 0.15% topical spray to suppress HPA axis function in patients with mild to moderate plaque psoriasis.
- 2. The secondary objectives are to evaluate the efficacy parameters and adverse event (AE) profile of desoximetasone 0.15% topical spray administered to patients with mild to moderate plaque psoriasis.

#### 9.0 INVESTIGATIONAL PLAN

## 9.1 Study Design and Plan Description

This open label, safety study is designed to evaluate the potential for adrenal suppression after treatment with desoximetasone 0.15% topical spray (Taro Pharmaceuticals, U.S.A.), for the treatment of mild to moderate plaque psoriasis.

Approximately 25 to 50 eligible patients with plaque psoriasis that satisfy all eligibility criteria will be enrolled into the study at Visit 1. Patients must be at least 2 years of age, overall in good health. They should have a current diagnosis of mild to moderate plaque psoriasis with IGA score of at least 2 or 3.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

Thirty (30) patients, stratified by age with a confirmed diagnosis of moderate to severe plaque psoriasis with:

Cohort 1 – 10-20 patients age 12-18 years of age with 5-10% BSA affected

Cohort 2 – 10-20 patients age 6-11 years of age with 5-10% BSA affected

Cohort 3 – 5-10 patients age 2-5 years of age with 5-10% BSA affected

Cohorts will be enrolled in sequential order. Each cohort will initiate enrollment once the previous cohort has reached the minimum number of patients and a safety analysis has been reviewed. Each cohort will be enrolled based on the availability of patients.

Each cohort will be reviewed for the potential of HPA axis suppression. If at least 50% of patients in each Cohort experience HPA axis suppression once the minimum number of patients has been enrolled and completed the cohort, enrollment for that cohort will be stopped and no further cohorts will be initiated. If at least 35% of patients have experienced HPA axis suppression across cohorts combined during the study, enrollment will be discontinued and no other cohorts will be initiated. Cohort 2 will not begin until safety data has been reviewed for Cohort 1. The same process will be followed for each Cohort until the study is complete.

The enrollment in the individual Cohort may not be required if the satisfactory safety data for the same age group was obtained in the study DSXS 1503.

Patients enrolled in the study will apply product twice a day, according to provided instructions, for a total of 28 days.

Patients will attend a total of 3 Clinic Visits as follows:

- Visit 1 (Day 1): Screening/Enrollment
- Visit 2 (Day  $14 \pm 2$ ): Interim Visit
- Visit 3 (Day  $29 \pm 2$ ): End of Study or Early Termination

The primary endpoint is the proportion of patients in the study with HPA axis suppression following treatment with the study medication.

The safety profile of each treatment group will be evaluated by comparing adverse events.

Ethical consideration related to this protocol and the use of human patients will be reviewed by an IRB.

# 9.2 Selection of Study Design

This open label, safety study to assess the potential of desoximetasone 0.15% topical spray to suppress HPA axis function was based on recommendations provided by the FDA in IND 101789 Guidance Meeting (01/14/2015, Reference ID 3689041), regarding the scope and design of studies for desoximetasone 0.15% spray and an FDA Advice Letter dated 04/27/2015. 10, 14

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# 9.3 Selection of Study Population

#### 9.3.1 Inclusion Criteria

- 1. Male or non pregnant, non lactating females:
  - **Cohort 1** 12-18 years of age
  - **Cohort 2** 6-11 years of age
  - Cohort 3 2-5 years of age
- 2. If female and of child bearing potential, have a negative urine pregnancy test at the baseline/ randomization visits and prepared to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g., condom with spermicide, IUD, oral, injected, transdermal or implanted hormonal contraceptives).
- 3. Signed informed consent form which meets all current ICH/FDA regulations. For patients under the age of majority in the state the study is being conducted (18 years in most states) the parent or legal guardian should sign the consent form and the child will be required to sign a patient "assent" form that will be written in such a way as to be understandable to a child.

Based on the patient's age 11 -17 years old will read and sign an IRB approved assent form. Patients 6-10 years of age will provide verbal assent to participate.

- 4. Patients with a definite clinical diagnosis of stable plaque psoriasis with involvement of:
  - Cohort 1 –age 12-18 years of age with 5-10% BSA affected (excluding face and scalp)
  - Cohort 2 –age 6-11 years of age with 5-10% BSA affected (excluding face and scalp)
  - Cohort 3 –age 2-5 years of age with 5-10% BSA affected (excluding face and scalp)
- 5. Investigator Global Assessment (IGA) score of 2 (mild) or 3 (moderate) at baseline (see Appendix B) for the overall disease severity.

## 9.3.2 Exclusion Criteria

- 1. Patients under 2 years of age.
- Females who are pregnant, lactating or likely to become pregnant during the study, or if of child bearing potential and sexually active not willing to use appropriate contraceptive methods to avoid pregnancy.
- 3. Plaque psoriasis with a BSA involvement of < 5% or > 10%.
- 4. Investigator Global Assessment (IGA) of less than 2 (mild) or greater than 3 (moderate) at baseline.
- 5. Current diagnosis of types of psoriasis other than stable plaque psoriasis (i.e., erythrodermic, exfolative or pustular psoriasis).
- 6. Patient who will require active treatment with a restricted medication during the study.
- 7. History of psoriasis that has been unresponsive to topical corticosteroid therapy.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

- 8. In the Investigator's opinion, the patient has other dermatological conditions, such as atopic or contact dermatitis, that may interfere with the clinical assessments of the signs and symptoms of psoriasis.
- 9. History of allergy or sensitivity to corticosteroids or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the patient or the results of the study.
- 10. History of an adverse reaction to Cortrosyn<sup>TM</sup> or similar test reagents.
- 11. Significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participation in the study.
- 12. Any radiation therapy, anti-neoplastic agents or immunosuppressant medication within 4 weeks before the first dose of study drug.
- 13. Treatment with any systemic antipsoriatic therapy or phototherapy (UVB or UVA) within 8 weeks before the first dose of study drug.
- 14. Treatment with any biological therapies for psoriasis within 12 weeks (or five half-lives whichever is less) before the first dose of study drug.
- 15. Treatment with any systemic steroids within 4 weeks of the first dose of the study drug. The use of inhaled or intranasal corticosteroids is acceptable as long as usage has been stable for at least 2 weeks before the first dose of study drug and will be continued during the study.
- 16. Use of any topical antipsoriatic agents of any kind or any topical corticosteroids for any reason within 2 weeks before first use of study drug. Nonprescription antipsoriatic shampoos used only on the scalp will be allowed during the study.
- 17. Inability to understand the protocol requirements, instructions, and study-related restrictions, the nature, scope, and possible consequences of the clinical study.
- 18. Unlikely to comply with the protocol requirements, instructions, and study-related restrictions, such as uncooperative attitude, inability to return for follow-up visits, and improbability of completing the clinical study.
- 19. Receipt of any drug as part of a research study within 30 days before first dosing.
- 20. The patient is a member of the investigational study staff or a member of the family of the investigational study staff.
- 22. Previous participation in this study including previous enrollment in DSXS 1503.

# 9.3.3 Restrictions during the Study

The following medications will not be allowed for the specified wash-out periods and throughout the study:

- Any prescription or over the counter (OTC) topical, systemic, phototherapy or biological medications for treatment of psoriasis.
- New regimens of anti-histamines

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

- O The use of anti-histamines, such as diphenhydramine, may be acceptable on condition that the patient has been on a stable dose for at least 14 days prior to enrollment and will remain on a stable dose throughout the study.
- Any oral, topical or injectable steroid drug use (with the exception of contraceptives).
  - Female patients using hormonal contraceptives should have been on the same product/dosing regimen for at least 28 days prior to and should not change this during the study.
- New regimens of inhaled corticosteroids.
  - o Inhaled corticosteroids are permissible, provided that the patient has been on a stable regimen for at least 2 weeks before the first dose of study drug and will continue during the study.
- Any other treatments, prescription or over the counter products for the treatment
  of any other dermatological condition including; topical corticosteroids,
  antibacterial, medicated and/or astringent washes, soaps, pads or moisturizers
  during the study.
- Use of high strength (20% or above) alpha-hydroxy acid or any kind of peel or other procedures on the treatment area during the study.

Patients and parents/legal guardians will be advised that the patient should avoid environmental conditions that may exacerbate their disease state such as excessive windy conditions and excessive exposure to sunlight. Patients and parents/legal guardians will be provided with a sunscreen for situations in which sun exposure cannot be avoided.

Patients and parents/legal guardians will be instructed not to apply the medication to the face, groin or axilla and not to use occlusive dressings on the treatment area.

Patients and parents/legal guardians will be questioned about all concomitant prescription and OTC medication use at each study visit. All concomitant medications (including use of the sunscreen if needed) will be recorded in the patient's study chart. Any patient or parents/legal guardians who violates any of the listed restrictions may be dropped from continued participation in the study by the Investigator.

# 9.3.4 Removal of Patients from the Study

Patients and parents/legal guardians will be advised that they are free to withdraw from the study at any time for any reason or, if necessary, the Investigator may withdraw a patient from the study to protect the health of that patient. A patient may also be withdrawn for not complying with study procedures. The clinical report will include all reasons for early withdrawals.

All patients who administer at least one dose of randomized study medication will be included in the safety analysis. If a patient terminates from the study early, all efforts will be made to complete their next visit study procedures. In case of early termination the Investigator shall fully document the reason for early termination. Reasons for early termination may include the following:

- Patient withdrew consent
- Significant adverse event that led the Investigator or patient to withdraw for safety reasons

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

- Worsening signs/symptoms
- Development of an intercurrent condition or complication that could affect the safety of the patient or the validity of the evaluation of the patient's clinical state to an extent considered significant by the Investigator
- Signs and symptoms of possible HPA axis suppression
- Protocol deviations/violations that in the Investigator's opinion warrant discontinuation

Non-compliance with dosing need not be a reason for early termination. Patients who withdraw or are removed from the study will not be replaced. In the event a patient withdraws or is dropped from the study for any reason, the Investigator will request return of the unused product and report the reason for the discontinued participation.

When a patient discontinues early from the study, all study procedures required for the end of study should be performed at their last study visit. Patients who are discontinued from the study after enrollment will be evaluated for safety and will be given, or referred for, appropriate treatment.

## 9.4 Treatments

#### 9.4.1 Treatments Administration

The patient or parent/legal guardian will be instructed to apply and rub in gently a thin film of the study drug to the affected areas twice daily (morning and evening) for 28 days. The hands should be washed after applying the drug.

To ensure compliance with the dosing technique, the patient or parent/legal guardian will be instructed to apply the first dose of medication under staff supervision at the time of enrollment and then twice daily until the patient's next scheduled visit. Patients and parents/legal guardians will be instructed not to apply the study drug within 12 hours of the visit which includes the Cortisol Response Test. Each patient or parent/legal guardian will be provided with a dosing diary in which they will be required to record dosing dates and times. These diaries should be brought to each visit in order that the study staff may check compliance. At the end of the study, the dosing diaries will be retained in the patient's file as source documentation.

At Visit 1 (Screening/Enrollment) and Visit 2 (Interim Visit) qualified study patients or parents/legal guardians will be provided with one 100 ml bottle of desoximetasone topical spray, 0.15% along with instructions for dosing. This bottle should be weighed before dispensing and the weight recorded. At Visit 2 (Interim Visit), the bottle should be collected, weighed and the weight recorded. A new 100 ml bottle of desoximetasone topical spray, 0.15% should be dispensed along with dosing instructions. The weight of the new bottle should be recorded before dispensing. This bottle will be returned and weighed at Visit 3 (End of Study/End of Treatment).

Treatment compliance will be encouraged by instructing the patient or parent/legal guardian on the proper dosing technique and by the use of the daily diary. Compliance will be assessed by evaluation of the diary.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# 9.4.2 Identity of Investigational Product

All study drugs will be provided by Taro Pharmaceuticals U.S.A., Inc. Each patient will receive 2 x 100 mL bottles of desoximetasone 0.15% topical spray.

The study medication will be shipped to each Investigator's site from a centralized pharmacy. The Principal Investigator at each site is responsible for ensuring that all study medications are stored in a locked, secure location, with access limited to the Investigator and his/her designee(s). An accurate inventory of the study medication will be maintained in accordance with federal regulations.

Once the site has been notified that they may do so, all unused study medication and empty or partially used bottles of study medication may be returned to the Sponsor or designee.

## 9.4.3 Method of Assigning Patients to Treatment Groups

Patients eligible for enrollment into the study will fall into one of four cohorts:

Cohort 1 – 10-20 patients age 12-18 years of age with 5-10% BSA affected

Cohort 2 – 10-20 patients age 6-11 years of age with 5-10% BSA affected

Cohort 3 – 5-10 patients age 2-5 years of age with 5-10% BSA affected

To ensure equivalent distribution of groups across sites Investigators will be required to contact Novum prior to enrollment.

At Visit 1 eligible patients will be enrolled to the study and assigned a patient number.

Cohorts will be enrolled in sequential order. Each cohort will initiate enrollment once the previous cohort has reached the minimum number of patients and a safety analysis has been reviewed. Each cohort will be enrolled based on the availability of patients.

Each cohort will be reviewed for the potential of HPA axis suppression. If at least 50% of patients in each Cohort experience HPA axis suppression once the minimum number of patients has been enrolled and completed the cohort, enrollment for that cohort will be stopped and no further cohorts will be initiated. If at least 35% of patients have experienced HPA axis suppression across cohorts combined during the study, enrollment will be discontinued and no other cohorts will be initiated. Cohort 2 will not begin until safety data has been reviewed for Cohort 1. The same process will be followed for each Cohort until the study is complete.

The enrollment in the individual Cohort may not be required if the satisfactory safety data for the same age group was obtained in the study DSXS 1503.

## 9.4.4 Packaging

This is an open label study. The study drug will contain a label with the following information:

- Protocol number
- Bottle number
- Space for patient number, patient's initials and dispensed date
- A note that the drug is for Investigational Use Only

# 9.4.5 Accountability

• The Investigator or designee will maintain an inventory of all study drug supplies received.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

- The Investigator or designee will maintain a log of all drug dispensed to and returned by the patients and note the date each drug is returned to the Sponsor.
- The weight of the study drug bottles before dispensing and after collection will be recorded.
- All study drug will be stored at controlled room temperature between 20°C to 25°C (68°F to 77°F), excursions permitted to 15°C to 30°C (59°F to 86°F), in a secure place with access to authorized individuals only.
- In the event of loss or apparent spoilage of the test preparation, the Investigator or designee must inform the study monitor. If necessary, a properly labeled replacement bottle will be issued to the patient.

# 9.4.6 Compliance

Patients will be provided with a diary with instructions to record the time and date of dosing. Patients will be asked to also record any adverse events and concomitant medications taken during the study.

Patients will dose twice daily for 28 days. All patients who are enrolled and used at least 75%-125% of scheduled doses of the study drug and have data from a post-treatment cortisol response test will be included in the analysis.

# 9.5 Study Conduct

The cortisol response test is to be done in the morning as the body's peak cortisol level is directly related to the event of awakening. Visit 1 and the Visit 3 should be scheduled before noon and subjects should not apply the study drug within 12 hours of Visit 3.

## 9.5.1 Visit 1 (Day 1): Screening/Enrollment, Before 12 pm

- 1. **Informed Consent:** For patients under the age of majority in the state the study is being conducted (18 years in most states) the parent or legal guardian should sign the consent form and the child will be required to sign a patient "assent" form that will be written in such a way as to be understandable to a child.
- 2. **Medical History and Demographics**: The patient's demographic and a complete medical history will be obtained for the patient's current and past medical conditions.
- 3. **Physical Examination and % BSA Assessment:** A general physical exam will be completed. The Subject's body weight (kg) and height (cm) will also be measured while the Subject is lightly clothed (e.g., no coat or shoes). %BSA will be assessed using instructions in Appendix A.
- 4. **Vital Signs:** The patient's vital signs will be recorded (pulse, blood pressure, temperature and respiration rate).
- 5. **Pregnancy Test:** A urine pregnancy test will be required of all women of child bearing potential prior to enrollment.
- 6. **IGA Score:** An investigator global assessment score will be completed. See Appendix B.
- 7. **Application Site Reactions:** Site of application will be assessed using instructions in Appendix C

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

- 8. **Concomitant Medication:** Review with the patient and parent/legal guardian the patient's use of concomitant medication within the last 12 weeks.
- 9. **Confirm Inclusion/Exclusion Met:** Confirm the patient meets all inclusion/exclusion criteria pending results of the Cortisol Response Test.
- 10. **Laboratory Evaluations:** A blood sample will be collected for hematology and clinical chemistry testing. (See Appendix F).
- 11. **Cortisol Response Test:** All patients will have a cortisol response test performed according to the procedure detailed in Appendix D.
- 12. **Dispense Study drug**: If patient is eligible to enroll, record the weight of one bottle of study drug and dispense with instructions.
- 13. **Apply Study Medication:** The first dose of study medication should be administered by the patient or parent/legal guardian at the site, under staff supervision.
- 14. **Provide Dosing Diary**: Provide Diary and instruct parent/legal guardian regarding how it is to be filled out and how study drug is to be used.
- 15. **Dispense Sunscreen:** For use only when sun exposure cannot be avoided.
- 16. **Provide Patient Wristband:** Each patient will receive a wristband to indicate that the patient is using a medication that has the potential to cause HPA axis suppression.
- 17. Schedule Visit 2.

## 9.5.2 Visit 2 (Day $14 \pm 2$ ): Interim Visit

- 1. **Pregnancy Test:** A urine pregnancy test will be required of all females of child bearing potential prior to enrollment.
- 2. **Vital Signs:** The patient's vital signs will be recorded (pulse, blood pressure, temperature and respiration rate).
- 3. **% BSA Assessment:** % BSA covered with plaque psoriasis will be assessed using instructions in Appendix A.
- 4. **IGA Score:** An investigator global assessment score will be completed. See Appendix B.
- 5. **Application Site Reactions:** Site of application will be assessed using instructions in Appendix C.
- 6. **Concomitant Medication:** Review with the patient and parent/legal guardian the patient's use of new or change in ongoing concomitant medication since Visit 1.
- 7. **Adverse Events:** Patients will be questioned about any health status changes/adverse events since last visit. All events will be recorded.
- 8. **Evaluation of Patient Compliance to the Protocol**: Collect and review patient's dosing diary for compliance and provide a new diary. Non-compliance with dosing does not warrant dismissal from the study. Counsel non-compliant patients and parents/legal guardians on dosing requirements of the study.
- 9. **Collect Study Drug:** The used bottle of study drug will be collected and the weight recorded.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

- 10. **Dispense Study drug**: If patient continues in the study, record weight of one bottle of study drug and dispense.
- 11. **Provide Dosing Diary:** If patient continues in the study, provide a new dosing diary. <u>Instruct parents/legal guardians not to apply dose to patient within approximately 12 hours of Visit 3.</u>

## 9.5.3 Visit 3 (Day $29 \pm 2$ ): End of Study or Early Termination, Before 12 pm

- 1. **Vital Signs:** The patient's vital signs will be recorded (pulse, blood pressure, temperature and respiration rate).
- 2. **Pregnancy Test:** A urine pregnancy test will be required of all women of child bearing potential prior to enrollment.
- 3. **Physical Exam:** A general physical exam will be conducted.
- 3. **% BSA Assessment:** % BSA covered with plaque psoriasis will be assessed using instructions in Appendix A.
- 4. **IGA Score:** An investigator global assessment score will be completed. See Appendix B.
- 5. **Application Site Reactions**: Site of application will be assessed using instructions in Appendix C.
- 6. **Concomitant Medication:** Review with the patient and parent/legal guardian the patient's use of new or change in ongoing concomitant medication since Visit 2.
- 7. **Adverse Events:** Patients will be questioned about any health status changes/adverse events since last visit. All events will be recorded.
- 8. **Evaluation of Patient Compliance to the Protocol**: Collect and review patient's dosing diary for compliance. Non-compliance with dosing does not warrant dismissal from the study. Counsel non-compliant patients and parents/legal guardians on dosing requirements of the study.
- 9. Collect Study Drug: The used bottle of study drug will be collected and the weight recorded.
- 10. **Laboratory Evaluations:** A blood sample will be collected for hematology and clinical chemistry testing. (See Appendix F)
- 11. **Cortisol Response Test:** All patients will have a cortisol response test performed according to the procedure detailed in Appendix D.

## 9.5.4 Visit 4 (Day $42 \pm 4$ ): Follow-up Phone Call

A phone call will be conducted approximately 14 days after the subject has completed dosing to follow-up on any new adverse events that may have occurred.

# 9.6 Study Procedures

# 9.6.1 Informed Consent

For patients under the age of majority in the state the study is being conducted (18 years in most states) the parent or legal guardian should sign the consent form and for patients 11 years of age or

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

older, an assent form will also be required. For illiterate parents or legal guardians, verbal consent should be obtained in the presence of and be countersigned by a literate witness. If any other language is required, translation will be performed by a certified translator. The child will be required to sign a patient "assent" form that will be written in such a way as to be understandable to a child. Patients 6-10 years of age will provide verbal assent to participate.

## 9.6.2 Demographics

At screening, each patient shall be required to provide basic demographic information: date of birth, gender, ethnicity and race.

# 9.6.3 Medical History

At Visit 1, patients will be questioned about medical history, including acute and chronic medical history and medical history relevant to their psoriasis, as well as all medication use within the past 12 weeks.

# 9.6.4 Vital Signs

The patient's vital signs will be recorded (heart rate, blood pressure, temperature and respiration rate) at Visit 1, 2, and 3.

# 9.6.5 Physical Exam and % Body Surface Area (BSA)

A general physical exam will be conducted at Visit 1 and Visit 3. At Visit 1 the patient's height (meters) and weight (kg) will be measured. The height and weight will be recorded and the Body Surface Area (BSA) will be calculated (see Appendix A for conversions from inches and pounds as appropriate). At Visits 1, 2 and 3, the % BSA affected will be recorded (see Appendix A).

## 9.6.6 Application Site Reaction Assessment

At Visits 1, 2 and 3, the application site reactions will be recorded (see Appendix C).

## 9.6.7 Investigator Global Assessment

At Visit 1 a visual inspection to confirm a diagnosis of chronic plaque psoriasis will be done. At each visit the Investigator will perform an Investigator Global Assessment (IGA) (See Appendix B). At Visit 1 the patient must have a IGA of 2 (mild) or 3 (moderate) for inclusion in the study.

## 9.6.8 Concomitant Medication Use

At Visits 1-3 patients will be questioned about current and concomitant medication use over the previous 12 weeks. At all visits patients will be questioned about ongoing or new concomitant medication use.

# 9.6.9 Pregnancy Test

Urine pregnancy tests on women of child-bearing potential will be performed at Visit 1, 2, and 3. The test must be negative for the patient to be eligible for inclusion in the study. If the patient is of non-childbearing potential, the source document must list the reason why she is of non-childbearing potential (e.g., premenarchal).

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

Any patient who becomes pregnant during the study must be discontinued and End of Study procedures completed. The outcome of the pregnancy will be followed by the Investigator to birth or early termination as appropriate. The pregnancy will be reported as an AE.

## 9.6.10 Dispensing Study Drug

At Visit 1 patients that satisfy all of the inclusion/exclusion criteria will be dispensed one bottle of the study drug and dosing instructions. At Visit 2 (Day 14) a new bottle of study drug will be dispensed.

The weight of the study drug product should be recorded before dispensing. The patient will be instructed to apply the first dose of study drug during Visit 1 under staff supervision.

## 9.6.11 Collecting Study Drug

Study medication bottles will be collected and weighted at Visits 2 and 3.

# 9.6.12 Dosing Instructions and Diary

Patients will be given a dosing diary and will be instructed on how to complete the diary. Patients will be asked to record the time and date of each dose, AEs, and concomitant medications throughout the study. The diary will be reviewed at each visit by the study staff.

## 9.6.13 Dosing Compliance

Dosing compliance will be checked by site staff at Visits 2 and 3. Patients taking fewer than 75% or more than 125% of the scheduled doses will be considered non-compliant with dosing. Compliance with dosing will be verified by the use of the patient diaries.

# 9.6.14 Standard Sunscreen and Patient Wristband

All patients will be advised to avoid sun exposure. A standard sunscreen will be provided at Visit 1 should the use of sunscreen be warranted. Each patient who enters the study will be provided with a wristband at Visit 1 to identify that the patient is taking a medication that could potentially cause HPA Axis Suppression. The patient should be instructed to wear the wristband for the duration of study.

# 9.6.15 Laboratory Evaluation

At Visit 1 and Visit 3 a blood sample will be collected for hematology and clinical chemistry testing (See Appendix E).

#### 9.6.16 Cortisol Response Test

At Visit 1 and Visit 3 all patients will have a cortisol response test performed according to the procedure detailed in Appendix E. The resulting blood sample should be sent to ACM Global Laboratory for immediate testing.

## Visit 3 Test

The test at the End of Study visit should not be performed if the patient dosed within 12 hours.

A patient will be considered to have normal basal cortisol level and adrenal function if they meet all three criteria listed below under Normal. Failure to meet any of these criteria is indicative of abnormal adrenal function or potential HPA axis suppression, even in absence of related symptoms

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

(e.g. nausea, headache, myalgia, fatigue or loose stool); in case of abnormal results, the patient will be monitored in accordance to the follow-up schedule below.

| | Cortisol Results | |
|---|---|---|
| | Normal | Abnormal |
| Basal | | |
| (pre Cortrosyn <sup>TM</sup> | $\geq 5 \text{ mcg/}100\text{ml}$ | < 5 mcg/100ml |
| injection) | _ | |
| 30 minutes post | ≥ basal value + 7 | < basal value + 7 |
| Cortrosyn <sup>TM</sup> injection | > 18 mcg/100ml | $\leq 18 \text{ mcg/}100\text{ml}$ |

HPA Axis suppression will be defined as a 30 minute post Cortrosyn<sup>TM</sup> injection level cortisol level of  $\leq$  18 mcg/100ml. As the study treatment period will be over, any patients with results of HPA axis suppression will be advised not to initiate any new steroid therapy, topical or otherwise, and to return to the site in 28 days at which time they will be assessed for HPA axis suppression.

Any patient presenting with symptoms of HPA axis suppression, such as nausea, headache, myalgia, fatigue or loose stool, will be referred to an endocrinologist. As an additional safety precaution, wristbands identifying the patient as someone suffering from adrenal suppression secondary to steroid withdrawal will be provided to alert medical personnel should any emergencies arise before adrenal function returns to normal.

If the results of the cortisol response test still show signs of HPA axis suppression 28 days after discontinuing therapy the patient will be asked to return in 28 days (56 days after discontinuing steroid therapy) for another follow-up test. If the patient is still showing signs of HPA axis suppression 56 days after discontinuing steroid therapy and presents with related symptoms, the patient will be referred to an endocrinologist.

If HPA axis suppression persists for 56 days after discontinuing steroid therapy, but the patient has no symptoms they will be asked to return in 28 days (84 days after discontinuing steroid therapy) for another follow-up test. If HPA axis suppression persists for 84 days after discontinuing steroid therapy the patient will be referred to an endocrinologist regardless of symptoms.

Patients should not be subjected to Cortrosyn<sup>TM</sup> testing, or any other challenge to their adrenal response, any sooner than 4 weeks from their last Cortrosyn<sup>TM</sup> test.

Follow-Up Schedule for Patients showing signs of HPA Axis Suppression

| Days | HPA Results | Symptoms | Patient Course |
|-----------|-------------|-----------|-----------------------------|
| after d/c | | | |
| 28 | Normal | N/A | Study over |
| 28 | Abnormal | Yes | Refer to endocrinologist |
| 28 | Abnormal | No | Repeat test in 28 days |
| 56 | Normal | N/A | Study over |
| 56 | Abnormal | Yes | Refer to endocrinologist |
| 56 | Abnormal | No | Repeat test in 28 days |
| 84 | Normal | N/A | Study over |
| 84 | Abnormal | Yes or No | Refer to an endocrinologist |

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

#### 9.7 Adverse Events

The patients will be monitored throughout the study for any Adverse Events (AEs). AEs will be collected through both solicited and unsolicited means and subsequently coded in tabular form using the MedDRA (Version 19 or higher) Adverse Event Dictionary. The patients will be encouraged to report signs, symptoms, and any changes in health to the clinic staff. Severity of each AE will be determined by the staff based on observation and questioning of the patients. The Investigator will judge the relationship of the event to the study treatments. Adverse events should be followed up until they have resolved or stabilized.

## 9.7.1 Adverse Event Definitions

Adverse Event: Any untoward medical occurrence in a patient or clinical investigation patient administered a pharmaceutical product and which does not necessarily have a causal relationship with treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease, temporally associated with the use of a medicinal (investigational) product, whether or not related to this product. This includes events not seen at baseline, or worsened even if present at baseline.

<u>Unexpected Adverse Event:</u> An adverse event where the nature or severity of is not consistent with the applicable product information (e.g., Investigator's Brochure for an unapproved investigational product or package insert/summary of product characteristics for an approved product).

Adverse Drug Reaction: All noxious and unintended responses to a medical product related to any dose should be considered adverse drug reactions. The response to a 'medical product' means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility, i.e., the relationship cannot be ruled out.

## 9.7.2 Severity of Adverse Event

The severity of the adverse event will be graded by the Investigator using the following criteria as guidelines:

- MILD: Awareness of symptom but does not interfere with routine activities.
- MODERATE: Discomfort sufficient to interfere with routine activities.
- SEVERE: Impossible to perform routine activities.

## 9.7.3 Relationship of Adverse Event

Relationship to the Study Product

- NOT RELATED: Any AE that is clearly not related to use of the study drug.
- POSSIBLE: The association of the AE with the study drug is unknown; however, a relationship between the drug and event cannot be ruled out.
- PROBABLE: There is reasonable temporal relationship between the use of the study drug and the AE. Based upon the Investigator's clinical experience, the association of the event with the study drug seems likely.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

DEFINITE: The AE occurs following the application of the study drug and it cannot be
reasonably explained by any other known characteristics of the patient's clinical state,
environmental or toxic factors, or other modes of treatment administered to the patient. It
disappears or decreases upon discontinuation of the study medication and reappears on a
re-challenge of the study drug.

# 9.7.4 Patient Participation Stopping Criteria

In the opinion of the Investigator, if the patient suffers an AE that warrants discontinuation of the study drug due to interference with age-appropriate instrumental ADL (Activities of Daily Living), for example preparing for meal, shopping for groceries or clothing, using the telephone, etc. the patient will be followed until the AE resolves or is considered stable. Any subject that discontinues the study due to an adverse event will be followed until resolution or stabilization of the adverse event.

#### 9.8 Serious Adverse Events

#### 9.8.1 Definition of a Serious Adverse Event

A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose suggests a medically significant hazard, including any event that:

- Results in death includes all deaths, even those that appear to be completely unrelated to study treatment (e.g., car accident where patient is a passenger).
- Is life—threatening in the view of the Investigator, the patient is at immediate risk of death at the time of the event.
- Results in persistent or significant disability or incapacity (substantial disruption of one's ability to conduct normal life).
- Requires inpatient hospitalization or prolongation of existing hospitalization.
- Causes congenital anomaly or birth defect.
- Is an important medical event that may not be immediately life-threatening or result in death or hospitalization, but may jeopardize the patient or may require medical or surgical intervention to prevent one of the serious outcomes listed above (e.g., intensive treatment in an emergency room, convulsions that do not result in hospitalizations). Emergency Room visits that require medical or surgical intervention to prevent one of the other serious outcomes listed above are considered a Serious Adverse Event.

## 9.8.2 Reporting Serious Adverse Events

# **Investigator Reporting of SAEs**

Adverse events which are evaluated by the Investigator as "Serious" will be reported to the Sponsor and IRB within 24 hours of notice whether or not they are considered expected or drug-related. All SAEs will be reported as per applicable regulations. All SAEs encountered during the study will be reported on the appropriate form and summarized in the final report.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# Any serious or unexpected adverse events should be reported to Novum within 24 hours. Following is the contact information:

Gail Gongas

Vice President, Clinical Trials Cell Phone 412-606-1603 Phone 412-363-3300 x 522 Fax 412-291-3171

-271-

Or

Paolo Fanzio, MD Medical Monitor Phone 412-363-3300 x 597 Fax 412-291-3171

Novum will report any Serious Adverse Event to Taro.

Documentation should be sent to Taro's Study Manager and/or Taro's Drug Safety Department listed below:

<u>Taro Study Manager:</u> <u>Taro Drug Safety Manager:</u>

Natalie Yantovskiy Margo Lacy Wyatt, RN, BSN,

Director, Clinical Research Associate Director, Drug Safety

Taro Pharmaceuticals U.S.A., Inc.

Medical Affairs

3 Skyline Drive Taro Pharmaceuticals U.S.A., Inc.

Hawthorne, NY 10532 3 Skyline Drive, Hawthorne, NY 10532

Phone: (914) 345-9001 x 6849 914-345-9001 Ext. 6758

Email: Natalie. Yantovskiy@Taro.com Email: Margo. Wyatt@taro.com

and TAROPVUS@TARO.com

Investigators will be informed of any SAEs reported at other study sites within 15 days from the initial report.

## 10.0 STATISTICAL METHODS

# 10.1 Statistical Plan

A Statistical Analysis Plan (SAP), detailing the intended statistical analysis of the study data, will be prepared as a separate document and finalized before database lock. Any deviation from the original statistical plan will be described and justified in the final report, as appropriate. The procedure for accounting for missing, unused and spurious data will be included in the Statistical Analysis Plan.

All statistical analysis will be conducted using SAS®, Version 9.4 or higher.

#### 10.1.1 Determination of Sample Size

The sample size of 30 patients, stratified by age and % BSA, was determined to be sufficient for this study.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

## 10.1.2 Baseline Comparability

Baseline comparability of the two groups will be assessed using appropriate statistical tests (e.g., one-way analysis of variance, Fisher's exact test, Cochran-Mantel-Haenszel test). The groups will be compared for basic demographics (age, gender, ethnicity and race), baseline IGA and baseline total BSA. Summary tables by group will be presented.

# 10.1.3 Safety Analysis of Potential HPA Axis Suppression

Dosing will be twice a day for 28 days excluding the doses prior to the Cortisol Response Test (54 applications). All patients who are enrolled, use at least 42 doses of the study drug and have data from a post-treatment cortisol response test will be included in the analysis. Patients who have not used 42 doses of the study drug will be excluded from the primary analysis of HPA axis suppression.

The primary analysis of interest is the proportion of patients in each group who are considered to have demonstrated possible HPA axis suppression following treatment with the study medication. As a secondary analysis of the data a logistic regression of the proportion of patients in the study with HPA axis suppression will be performed with %BSA affected as a covariate. See Appendix D for results from the cortisol response test considered indicative of potential HPA axis suppression.

Cohorts will be enrolled in sequential order. Each cohort will initiate enrollment once the previous cohort has reached the minimum number of patients and a safety analysis has been reviewed. Each cohort will be enrolled based on the availability of patients.

Each cohort will be reviewed for the potential of HPA axis suppression. If at least 50% of patients in each Cohort experience HPA axis suppression once the minimum number of patients has been enrolled and completed the cohort, enrollment for that cohort will be stopped and no further cohorts will be initiated. If at least 35% of patients have experienced HPA axis suppression across cohorts combined during the study, enrollment will be discontinued and no other cohorts will be initiated. Cohort 2 will not begin until safety data has been reviewed for Cohort 1. The same process will be followed for each Cohort until the study is complete.

For all patients the actual amount of desoximetasone (mg) applied during the study will be calculated from recorded bottle weights and presented.

# 10.2 Safety Analysis

Safety analysis will be conducted on all patients who applied at least one dose of study drug.

Adverse medical events experienced by the patients will be tabulated. The relationship of AEs, if any, to the study drug will be assessed by the Investigator. Adverse events assessed as definite, probable, possible or not related to the study drug will be presented. Shift analysis using the categories; below, above and within the laboratory normal range will be performed to identify any specific laboratory parameter that shows a trend toward potentially clinically significant changes.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

## 11.0 REGULATORY OBLIGATIONS

#### 11.1 Institutional Review Board

The study protocol, informed consent/assent form, Investigator's Brochure, or package insert (as applicable), and any specific advertising will be submitted to, and approved by, an Institutional Review Board (IRB) before the start of the study. A form must be signed by the chairman or designee of the IRB noting the approvals. This notification of the board's approval along with a description by profession and gender of the board's composition will be provided to the Sponsor.

## 11.2 Study Documentation

This study will be conducted in compliance with the protocol, Good Clinical Practices (GCPs) and all applicable regulations, including the Federal Food, Drug and Cosmetics Act, US applicable Code of Federal Regulations (title 21), parts 50, 56, 312, 320 and any IRB requirements relative to clinical studies and the Declaration of Helsinki, June 1964, as modified by the 59<sup>th</sup> World Medical Association General Assembly, October 2013.

The Investigator will permit trial-related monitoring, audits, IRB review and regulatory inspections providing direct access to source data/documents.

## 11.2.1 Protocol

The Investigator indicated on FDA Form 1572 will act as the Principal Investigator at each study site. Protocols will be noted as approved by placement of the Novum Representative's signature on the cover page. The Sponsor of the study will also approve the protocol by having a study-responsible individual sign the protocol cover page.

#### 11.2.2 Informed Consent

An Informed Consent Form (ICF) that includes all of the relevant elements currently required by FDA and local State regulations will be provided to each prospective study patient's parent/legal guardian before enrollment into the study. In addition, subjects 11-17 years of age will be presented with an Assent Form. The type and method of study, tests to be administered, any potential or possible hazards, and the patient's right to withdraw from the study at any time will be explained to the patients by the Investigator or designee. Once the Investigator or designee is assured that an individual candidate understands the implications of participating in this study, the parent/legal guardian will be asked to give consent by signing and dating the ICF/Assent Form and the patient will be asked to give assent by signing and dating in the appropriate areas of the Assent. The Investigator or designee will also sign and date the form, along with a staff member who will sign the ICF as a witness to verify that the patient has indeed received information. For illiterate patients, verbal consent should be obtained in the presence of and be countersigned by a literate witness. If any other language is required, translation will be performed by a certified translator. A copy of the ICF will be provided to the patient.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

## 11.2.3 Protocol and Informed Consent Changes

Revisions to the original protocol will be documented in amendments, incorporated as a preface to the new version and approved by the IRB. Any revision that substantially alters the study design or increases potential risk to the patient requires the patient's consent to continue in the study. Revisions to the original ICF will also be approved by the IRB. The approvals will be processed in accordance with the established IRB procedures. Copies of all protocol and ICF amendments/revisions, along with letters noting IRB approval, will be submitted to the Sponsor.

## 11.2.4 Source Documents and Case Report Forms

All patients will be identified by initials, date of birth, and a unique patient number. Source documents will be used to record all study-related data. Source document entries will be used to complete Case Report Forms (CRFs). A set of CRFs will be completed for each patient enrolled in the study. All data and CRFs will be reviewed, evaluated and signed by the Investigator, as required.

The original source documents and a copy of the corresponding CRFs will be retained by the Investigator. Patients who terminate early from the study will have the end of study (Visit 3) source/CRF completed.

## 11.2.5 Drug Accountability

All drug receipt, inventory, dispensing, dosing and reconciliation records will be maintained in compliance with Federal Regulations. The study drug will be dispensed to qualified study patients according to established procedures. At the end of the study (after the database has been locked) all used and unused study drug will be returned to Novum.

## 11.2.6 Drug Storage

All study drug will be stored at controlled room temperature 15-30°C (59-86°F), in a secure place with access by authorized individuals only. The Investigator will be responsible for maintaining accurate records of drug receipt, dispensing, and return. At the end of the study, all partially used and unused study drug will be returned to Novum.

## 11.2.7 Pregnancies

Patients with a positive pregnancy test during screening will not be enrolled in the study. Patients who report that they have become pregnant during the study or have a positive pregnancy test at any clinic visit will be followed to completion of the pregnancy. The pregnancy will be reported as an AE.

Female patients of childbearing potential must have been using and must agree to continue to use accepted methods of birth control, throughout the study. All female patients are considered to be of childbearing potential unless they are premenarchal, have been surgically sterilized or have been postmenopausal for at least 1 year. Abstinence is an accepted method of birth control. Alternatively, any of the following methods of birth control are acceptable: oral contraceptives, contraceptive patches/implants (e.g., Norplant®), Depo-Provera®, double barrier methods (e.g., condom and spermicide) or IUD. Prior to study enrollment women of child bearing potential must be advised of the importance of avoiding pregnancy during study participation.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

A negative result of a urine pregnancy test having a minimum sensitivity of at least 25 mIU/ml for hCG should be obtained, prior to study participation. Pregnancy testing will be performed at Visits 1, 2, and 3 and the results of all pregnancy tests (positive or negative) will be documented.

If following initiation of study treatment, it is subsequently discovered that a study patient is pregnant or may have been pregnant at the time of Investigational Product exposure, the Investigational Product will be permanently discontinued. The Principal Investigator must immediately notify the Medical Monitor of this event.

Protocol-required procedures for study discontinuation and follow-up must be performed on the patient. Other appropriate pregnancy follow-up procedures should be considered if indicated. In addition, the Principal Investigator must report to the sponsor follow-up information regarding the course of the pregnancy, including perinatal and neonatal outcome. Infants should be followed for a minimum of eight weeks after birth.

# 11.2.8 Reporting Safety Information to the IRB

The Investigator must promptly report to the Investigator's IRB all unanticipated problems involving risks to patients. This includes death from any cause and all serious adverse events occurring during the study, regardless of the assessed causality.

#### 11.2.9 Record Retention

All drug accountability records, CRFs, source data and related regulatory documents must be retained for at least ten years following completion of the study or for two years after the test product has been approved for marketing by the Food and Drug Administration.

# 11.2.10 Study Monitoring and Auditing

Novum will be responsible for monitoring the study according to Good Clinical Practice and applicable regulations. Monitoring visits are for the purpose of confirming adherence to the protocol and to verify complete and accurate data collection. The clinical site will make all records associated with the study available to Novum's representative during such visits and audits

The study may be subject to audit by the Sponsor, Sponsor Representative or by regulatory authorities. If such an audit occurs the Investigator must agree to allow access to required patient records. By signing this protocol, the Investigator grants permission to personnel from the Sponsor, its representatives and appropriate regulatory authorities for on-site monitoring of all appropriate study documentation, as well as on-site review of study procedures.

#### 11.2.11 End of the Trial

The end of the trial is defined as the time at which the last patient has completed their last visit in the study. Upon completion of the study, the study drug will no longer be available to the patient but the Investigator can, at their discretion, discuss alternative treatments with the patient.
An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# 11.2.12 Clinical Study Report

At the end of the study a full report in e-CTD format will be prepared that will include a narrative of the clinical conduct and results of the study, a statistical report including a description of the analysis performed, and other documentation as may be appropriate.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

## 12.0 REFERENCES

- 1 <u>www.psoriasis.org</u>
- 2 Raychaudhuri SP, Gross J. A comparative study of pediatric onset psoriasis with adult onset psoriasis. Pediatr Dermatol. 2000;17(3):174-178.
- Augustin M, Glaeske G, Radtke MA, Christophers E, Reich K, Schafer I. Epidemiology and comorbidity of psoriasis in children. Br J Dermatol. 2010;162(3):633-636.
- 4 NDA#020-934. Connetics February 1999.
- Hengge UR, Ruzicak T, Schwartz RA, Cork MJ Adverse effects of Topical Glucocorticosteroids. J Am Acad Dermatology 2006 54:1 Continuing Medical Education.
- 6 Product Label for TOPICORT® (desoximetasone) Topical Spray, 0.25%, April 2013
- 7 Product Label for Cortrosyn TM Amphastar Pharmaceuticals, Inc. August 2009.
- 8 Summary Basis of Approval OLUX® clobetasol 0.05% foam. NDA#021-142. Connetics May 2000.
- 9 Summary Basis of Approval LUXIQ® betamethasone 0.12% foam.
- FDA Correspondence Meeting Minutes. IND 101789, Desoximetasone Topical Spray, 0.25%. Department of Health and Human Services, FDA 01/14/2015.
- Pediatric Burns. Physical Medicine and Rehabilitation Board Review. Cuccurullo S, editor. New York: Demos Medical Publishing; 2004.
- Thomas CL, Finlay AY. The 'handprint' approximates to 1% of the total body surface area whereas the 'palm minus the fingers' does not. Br J Dermatol 2007; 157(5): 1080-1.
- Mosteller RB. Simplified Calculation of Body Surface Area. N. Eng. J. Med. 1987; Oct 22 317(77): 1098
- FDA Correspondence Advice Letter. IND 101789. Department of Health and Human Services, FDA 04/27/2015.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

## 13.0 APPENDICES

## **APPENDIX A: Body Surface Area Calculation**

## **Total Body Surface Area Calculation**

To calculate the Total BSA the following procedure (Mosteller Formula<sup>13</sup>) should be followed.

Total Body Surface Area (BSA) in meters squared

 $m^2 = ((height (cm) x weight (kg)) / 3600)^{1/2}$ 

It is preferable that the patient's height and weight be measured in cm and kg however if needed:

To convert inches (in) to centimeters (cm) the following conversion should be used

1 inch = 2.54 cm

To convert pounds (lbs) to kilograms (kg) the following conversion should be used

1 lb = 0.45 kg

The patient's height and weight should be reported to the nearest cm and nearest 0.5 kg. The BSA should be reported to the nearest second decimal place.

For example a patient who is 68 inches tall and weighs 180 lbs will have a reported BSA of:

```
180 lb x 0.45 = 81.0 \text{ kg}

BSA = SQRT ((173 x 81.0)/3600)

= 1.97 m<sup>2</sup>
```

 $68 \text{ in } \times 2.54 = 173 \text{ cm}$ 

## **%BSA Affected**

To estimate the % BSA Affected, the Investigator should use the method of approximation:

The "Rule of Nines" provides a general estimation of total BSA for several anatomic areas (each arm = 9%, each leg = 18%, back = 18%, chest and abdomen = 18%, head = 9%, groin = 1%). The Investigator may then visually estimate the proportion of the involved skin within each anatomic area and calculate the total percentage of BSA affected. In children, hips and legs are smaller and the head, neck and shoulders are larger, as a result, a modified "Rule of Nines" is used (see diagram below).

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

| Part | 1-4 year child<br>body<br>% of total | 5-9 year child<br>body<br>% of total | 10-14 year child<br>body<br>% of total | 15 year-adult<br>body<br>% of total |
|---|---|---|---|---|
| Arm | 9.5% | 9.5% | 9.5% | 9% |
| Head | 19% | 15% | 12% | 9% |
| Neck | 19% | 13% | 1% | 1% |
| Leg | 15% | 17% | 18% | 18% |
| Anterior trunk | 16% | 16% | 16% | 18% |
| Posterior trunk | 16% | 16% | 16% | 18% |



An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# **APPENDIX B: Investigator Global Assessment (IGA)**

To be eligible for inclusion in the study the IGA must be 2 - 3 at baseline.

| Score | Category | Description |
|---|---|---|
| 0 | Clear | Plaque: elevation: no evidence of plaque elevation above normal skin level. |
| | | Scaling: no evidence of scaling |
| | | Erythema: no redness |
| 1 | Minimal | Plaque elevation: very slight elevation above normal skin level, easier felt than |
| | | seen |
| | | Scaling: limited amount of very fine scales partially covers some of the plaques |
| | | Erythema: very few of the plaques are light red |
| 2 | Mild | Plaque elevation: slight but definite elevation above the normal skin level, |
| | | typically with edges that are indistinct or sloped on some of the plaques. |
| | | Scaling: mainly fine scales, some plaques are partially covered. |
| | | Erythema: some plaques are light red |
| 3 | Moderate | Plaque elevation: moderate elevation with rounded or sloped edges on most of |
| | | the plaques |
| | | Scaling: somewhat coarser scales; most plaques are partially covered. |
| | | Erythema: most plaques are red |
| 4 | Severe | Plaque elevation: marked to very marked elevation, with hard to very hard sharp |
| | | edges on virtually all or all of the plaques. |
| | | Scaling: coarse, thick scales; virtually all or all plaques are covered; rough |
| | | surface. |
| | | Erythema: virtually all or all plaques are bright to dusky red. |

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# **APPENDIX C: Application Site Reactions**

| The following a | nnlication | site reactions | will be | evaluated a | t each visit | based or | n the scale | provided below: |
|---|---|---|---|---|---|---|---|---|
| ine rome wing a | ppiication | bite reactions | , ,,,,,,, | c raraatea a | t cacii vibit | oused of | ii tiic beare | provided below. |

| Burning | | |
|----------|---|------------------------------|
| Erosion | | |
| Edema | | |
| Pain | | |
| Itching | | |
| Dryness | | |
| Absent | 0 | |
| Mild | 1 | (slight, barely perceptible) |
| Moderate | 2 | (distinct presence) |
| Severe | 3 | (marked, intense) |

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

## **APPENDIX D: Cortisol Response Test**

This cortisol release test is modified from the procedure of Wood et al as described in the Product Label for Cortrosyn<sup>TM</sup> (cosyntropin) for injection (Amphstar Pharmaceuticals, Inc.).

The procedure is as follows:

- 1. A single 3 ml blood sample should be taken as the basal sample.
- 2. 0.25 mg (a single vial) of Cortrosyn<sup>TM</sup> (cosyntropin) should be reconstituted with 1.0ml of 0.9% sodium chloride injection USP injected intramuscularly. In patients under 3 years of age, 0.125mg of Cortrosyn<sup>TM</sup> will be used.
- 3. 30 minutes after the IM injection a second 3 ml blood sample should be obtained. The resulting two serum samples (at least 1 ml of serum in each) should be processed and labeled according to the instructions provided and sent the same day to ACM Global Laboratory for analysis of basal and post stimulated serum cortisol concentration.

At Visit 1 and Visit 3 all patients will have a cortisol response test performed according to the procedure detailed in Appendix C. The resulting blood sample should be sent to ACM Global Laboratory for immediate testing.

## Visit 1 Test

A cortisol response test will be conducted at Visit 1.

## Visit 3 Test

The test at the End of Study visit should not be performed if the patient dosed within 12 hours.

A patient will be considered to have normal basal cortisol level and adrenal function if they meet all three criteria listed below under Normal. Failure to meet any of these criteria is indicative of abnormal adrenal function or potential HPA axis suppression.

| | Cortisol Results | |
|---|---|---|
| | Normal | Abnormal |
| Basal (pre Cortrosyn <sup>TM</sup> injection) | ≥ 5 mcg/100ml | < 5 mcg/100ml |
| 30 minutes post | ≥ basal value + 7 | < basal value + 7 |
| Cortrosyn <sup>TM</sup> injection | > 18 mcg/100ml | $\leq 18 \text{ mcg/}100\text{ml}$ |

HPA Axis suppression will be defined as a 30 minute post Cortrosyn<sup>TM</sup> injection level cortisol level of  $\leq$  18 mcg/100ml. As the study treatment period will be over, any patients with results of HPA axis suppression will be advised not to initiate any new steroid therapy, topical or otherwise, and to return to the site in 28 days at which time they will be assessed for HPA axis suppression.

Any patient presenting with symptoms of HPA axis suppression, such as nausea, headache, myalgia, fatigue or loose stool, will be referred to an endocrinologist. As an additional safety precaution, wristbands identifying the patient as someone suffering from adrenal suppression secondary to steroid withdrawal will be provided to alert medical personnel should any emergencies arise before adrenal function returns to normal.

If the results of the cortisol response test still show signs of HPA axis suppression 28 days after discontinuing therapy the patient will be asked to return in 28 days (56 days after discontinuing steroid therapy) for another follow-up test. If the patient is still showing signs of HPA axis suppression 56 days

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

after discontinuing steroid therapy and presents with related symptoms, the patient will be referred to an endocrinologist.

If HPA axis suppression persists for 56 days after discontinuing steroid therapy, but the patient has no symptoms they will be asked to return in 28 days (84 days after discontinuing steroid therapy) for another follow-up test. If HPA axis suppression persists for 84 days after discontinuing steroid therapy patients will be referred to an endocrinologist regardless of symptoms.

Patients should not be subjected to Cortrosyn<sup>TM</sup> testing, or any other challenge to their adrenal response, any sooner than 4 weeks from their last Cortrosyn<sup>TM</sup> test.

Follow-Up Schedule for Patients showing signs of HPA Axis Suppression

| Days | HPA Results | Symptoms | Patient Course |
|-----------|-------------|-----------|-----------------------------|
| after d/c | | | |
| 28 | Normal | N/A | Study over |
| 28 | Abnormal | Yes | Refer to endocrinologist |
| 28 | Abnormal | No | Repeat test in 28 days |
| 56 | Normal | N/A | Study over |
| 56 | Abnormal | Yes | Refer to endocrinologist |
| 56 | Abnormal | No | Repeat test in 28 days |
| 84 | Normal | N/A | Study over |
| 84 | Abnormal | Yes or No | Refer to an endocrinologist |

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# APPENDIX E: Evaluation of HPA Axis Suppression Corticosteroid Effect on HPA Axis Feedback Loop



The Hypothalamus secretes Corticotrophin Releasing Hormone (CRH) which triggers the anterior pituitary to release Adrenocorticotrophin Hormone (ACTH). ACTH stimulates the adrenal cortex to release glucocorticosteroids into the bloodstream. Increased levels of circulating glucocorticoids in the bloodstream send a signal to the hypothalamus to decrease the secretion of CRH and also to the anterior pituitary to decrease the secretion of ACTH resulting in a decrease in circulating glucocorticosteroids. Exogenous corticosteroids, including those absorbed systemically through the skin, may also impart a message to the hypothalamus and anterior pituitary to decrease secretion of hormones. This may result in decreased circulating glucocorticosteroids and thus, a decreased response to glucocorticosteroids.

## Assessment of Corticosteroid Effect on HPA Axis Feedback Loop



Low circulating cortisol levels or a decreased response to cortisol are indicative of suppression of the activity of the HPA axis. In order to evaluate the HPA axis function of patients in this study, basal levels of cortisol in the blood will be measured at the end of treatment. Patients will then be injected with Cortosyn<sup>TM</sup>, a synthetic subunit of ACTH. Systemic administration of a synthetic subunit of ACTH should stimulate the Adrenal Cortex to release glucocorticosteroids, unless the patient has increased circulating levels of glucocorticosteroids for some time and the HPA axis has been suppressed. After 30 minutes have passed blood levels of cortisol will be measured again. Lack of, or limited release of glucocorticosteroids into the blood stream in response to the Cortosyn<sup>TM</sup> will administered indicate suppression of HPA axis function.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

## **APPENDIX F: Clinical Laboratory Testing**

As part of the Screening Procedures and at Visit 3 (or early termination for randomized patients only) patients will have a blood sample taken for hematology and clinical chemistry testing. The testing panel should include as a minimum the following tests:

## Hematology

- Hematocrit
- White blood cell count
- Platelets
- Hemoglobin
- Red blood cell count
- Differential white cell count

## Chemistry

- Alkaline phosphatase
- Total bilirubin
- Alanine transaminase
- Creatinine
- Aspartate transaminase
- Glucose
- Blood urea nitrogen

Clinical Laboratory Testing will be performed at a Central Laboratory

# **ACM Medical Lab, Inc.**

160 Elmgrove Park Rochester, NY 14624, USA

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# APPENDIX G: Cortrosyn<sup>TM</sup> Package Insert

# FOR DIAGNOSTIC USE ONLY CORTROSYN™

(cosyntropin) for Injection

#### DESCRIPTION

CORTROSYNTM (cosyntropin) for Injection is a sterile lyophilized powder in vials containing 0.25 mg of CORTROSYNTM and 10 mg of mannitol to be reconstituted with 1 mL of 0.9% Sodium Chloride Injection, USP. Administration is by intravenous or intramuscular injection. Cosyntropin is  $\alpha$  1 - 24 corticotropin, a synthetic subunit of ACTH. It is an open chain polypeptide containing, from the N terminus, the first 24 of the 39 amino acids of natural ACTH. The sequence of amino acids in the 1 - 24 compound is as follows:

#### CLINICAL PHARMACOLOGY

CORTROSYNTM (cosyntropin) for Injection exhibits the full corticosteroidogenic activity of natural ACTH. Various studies have shown that the biologic activity of ACTH resides in the N-terminal portion of the molecule and that the 1 - 20 amino acid residue is the minimal sequence retaining full activity. Partial or complete loss of activity is noted with progressive shortening of the chain beyond 20 amino acid residues. For example, the decrement from 20 to 19 results in a 70% loss of potency.

The pharmacologic profile of CORTROSYNTM is similar to that of purified natural ACTH. It has been established that 0.25 mg of CORTROSYNTM will stimulate the adrenal cortex maximally and to the same extent as 25 units of natural ACTH. This dose of CORTROSYNTM will produce maximal secretion of 17-OH corticosteroids. 17- ketosteroids and / or 17 - ketogenic steroids.

The extra-adrenal effects which natural ACTH and CORTROSYNTM have in common include increased melanotropic activity, increased growth hormone secretion and an adipokinetic effect. These are considered to be without physiological or clinical significance.

Animal, human and synthetic ACTH (1-39) which all contain 39 amino acids exhibit similar immunologic activity. This activity resides in the C-terminal portion of the molecule and the 22-39 amino acid residues exhibit the greatest degree of antigenicity. In contrast, synthetic polypeptides containing 1-19 or fewer amino acids have no detectable immunologic activity. Those containing 1-26, 1-24 or 1-23 amino acids have very little immunologic although full biologic activity. This property of CORTROSYNTM assumes added importance in view of the known antigenicity of natural ACTH.

#### INDICATIONS AND USAGE

CORTROSYNTM (cosyntropin) for Injection is intended for use as a diagnostic agent in the screening of patients presumed to have adrenocortical insufficiency. Because of its rapid effect on the adrenal cortex it may be utilized to perform a 30-minute test of adrenal function (plasma cortisol response) as an office or outpatient procedure, using only 2 venipunctures (see DOSAGE AND ADMINISTRATION section).

Severe hypofunction of the pituitary - adrenal axis is usually associated with subnormal plasma cortisol values but a low basal level is not per se evidence of adrenal insufficiency and does not suffice to make the diagnosis. Many patients with proven insufficiency will have normal basal levels and will develop signs of insufficiency only when stressed. For this reason a criterion which should be used in establishing the diagnosis is the failure to respond to adequate corticotropin stimulation. When presumptive adrenal insufficiency is diagnosed by a subnormal CORTROSYNTM test, further studies are indicated to determine if it is primary or secondary.

Primary adrenal insufficiency (Addison's disease) is the result of an intrinsic disease process, such as tuberculosis within the gland. The production of adrenocortical hormones is deficient despite high ACTH levels (feedback mechanism). Secondary or relative insufficiency arises as the result of defective production of ACTH leading in turn to disuse atrophy of the adrenal cortex. It is commonly seen, for example, as result of corticosteroid therapy, Sheehan's syndrome and pituitary tumors or ablation.

The differentiation of both types is based on the premise that a primarily defective gland cannot be stimulated by ACTH whereas a secondarily defective gland is potentially functional and will respond to adequate stimulation with ACTH. Patients selected for further study as the result of a subnormal CORTROSYNTM test should be given a 3 or 4 day course of treatment with Repository Corticotropin Injection USP and then retested. Suggested doses are 40 USP units twice daily for 4 days or 60 USP units twice daily for 3 days. Under these conditions little or no increase in plasma cortisol levels will be seen in Addison's disease whereas higher or even normal levels will be seen in cases with secondary adrenal insufficiency.

#### CONTRAINDICATION

The only contraindication to CORTROSYNTM (cosyntropin) for Injection is a history of a previous adverse reaction to it.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

#### **PRECAUTIONS**

#### General

CORTROSYNTM (cosyntropin) for Injection exhibits slight immunologic activity, does not contain animal protein and is therefore less risky to use than natural ACTH. Patients known to be sensitized to natural ACTH with markedly positive skin tests will, with few exceptions, react negatively when tested intradermally with CORTROSYNTM. Most patients with a history of a previous hypersensitivity reaction to natural ACTH or a pre-existing allergic disease will tolerate CORTROSYNTM. Despite this however, CORTROSYNTM is not completely devoid of immunologic activity and hypersensitivity reactions including rare anaphylaxis are possible. Therefore, the physician should be prepared, prior to injection, to treat any possible acute hypersensitivity reaction.

#### **Drug Interactions**

Corticotropin may accentuate the electrolyte loss associated with diuretic therapy.

#### Carcinogenesis, Mutagenesis, Impairment of Fertility

Long term studies in animals have not been performed to evaluate carcinogenic or mutagenic potential or impairment of fertility. A study in rats noted inhibition of reproductive function like natural ACTH.

#### Pregnancy

Pregnancy Category C. Animal reproduction studies have not been conducted with CORTROSYNTM (cosyntropin) for Injection. It is also not known whether CORTROSYNTM can cause fetal harm when administered to a pregnant woman or can affect reproduction capacity. CORTROSYNTM should be given to a pregnant woman only if clearly needed.

#### **Nursing Mothers**

It is not known whether this drug is excreted in human milk. Because many drugs are excreted in human milk, caution should be exercised when CORTROSYNTM (cosyntropin) for Injection is administered to a nursing woman.

#### Pediatric Use

(See DOSAGE AND ADMINISTRATION section.)

#### ADVERSE REACTIONS

Since CORTROSYNTM (cosyntropin) for Injection is intended for diagnostic and not therapeutic use, adverse reactions other than a rare hypersensitivity reaction are not anticipated. A rare hypersensitivity reaction usually associated with a pre-existing allergic disease and/or a previous reaction to natural ACTH is possible. Symptoms may include slight whealing with splotchy erythema at the injection site. There have been rare reports of anaphylactic reaction. The following adverse reactions have been reported in patients after the administration of CORTROSYNTM and the association has been neither confirmed nor refuted:

- bradycardia
- tachycardia
- hypertension
- peripheral edema
- rash

## DOSAGE AND ADMINISTRATION

CORTROSYNTM (cosyntropin) for Injection may be administered intramuscularly or as a direct intravenous injection when used as a rapid screening test of adrenal function. It may also be given as an intravenous infusion over a 4 to 8 hour period to provide a greater stimulus to the adrenal glands. Doses of CORTROSYNTM 0.25 to 0.75 mg have been used in clinical studies and a maximal response noted with the smallest dose.

A suggested method for a rapid screening test of adrenal function has been described by Wood and Associates (1). A control blood sample of 6 to 7 mL is collected in a heparinized tube. Reconstitute 0.25 mg of CORTROSYNTM with 1mL of 0.9% Sodium Chloride Injection, USP and inject intramuscularly. The reconstituted drug product should be inspected visually for particulate matter and discoloration prior to injection. Reconstituted CORTROSYNTM should not be retained. In the pediatric population, aged 2 years or less, a dose of 0.125 mg will often suffice. A second blood sample is collected exactly 30 minutes later. Both blood samples should be refrigerated until sent to the laboratory for determination of the plasma cortisol response by some appropriate method. If it is not possible to send them to the laboratory or perform the fluorimetric procedure within 12 hours, then the plasma should be separated and refrigerated or frozen according to need.

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

Two alternative methods of administration are intravenous injection and infusion. CORTROSYNTM can be injected intravenously in 2 to 5 mL of saline over a 2-minute period. When given as an intravenous infusion: CORTROSYNTM, 0.25 mg may be added to glucose or saline solutions and given at the rate of approximately 40 micrograms per hour over a 6-hour period. It should not be added to blood or plasma as it is apt to be inactivated by enzymes. Adrenal response may be measured in the usual manner by determining urinary steroid excretion before and after treatment or by measuring plasma cortisol levels before and at the end of the infusion. The latter is preferable because the urinary steroid excretion does not always accurately reflect the adrenal or plasma cortisol response to ACTH.

The usual normal response in most cases is an approximate doubling of the basal level, provided that the basal level does not exceed the normal range. Patients receiving cortisone, hydrocortisone or spironolactone should omit their pre-test doses on the day selected for testing. Patients taking inadvertent doses of cortisone or hydrocortisone on the test day and patients taking spironolactone or women taking drugs which contain estrogen may exhibit abnormally high basal plasma cortisol levels

A paradoxical response may be noted in the cortisone or hydrocortisone group as seen in a decrease in plasma cortisol values following a stimulating dose of CORTROSYNTM.

In the spironolactone or estrogen group only a normal incremental response is to be expected. Many patients with normal adrenal function, however, do not respond to the expected degree so that the following criteria have been established to denote a normal response:

- 1. The control plasma cortisol level should exceed 5 micrograms/100 mL.
- 2. The 30-minute level should show an increment of at least 7 micrograms/100 mL above the basal level.
- 3. The 30-minute level should exceed 18 micrograms/100 mL. Comparable figures have been reported by Greig and co-workers (2).

Plasma cortisol levels usually peak about 45 to 60 minutes after an injection of CORTROSYNTM and some prefer the 60-minute interval for testing for this reason. While it is true that the 60-minute values are usually higher than the 30-minute values, the difference may not be significant enough in most cases to outweigh the disadvantage of a longer testing period. If the 60-minute test period is used, the criterion for a normal response is an approximate doubling of the basal plasma cortisol value.

In patients with a raised plasma bilirubin or in patients where the plasma contains free hemoglobin, falsely high fluorescence measurements will result. The test may be performed at any time during the day but because of the physiological diurnal variation of plasma cortisol the criteria listed by Wood cannot apply. It has been shown that basal plasma cortisol levels and the post CORTROSYNTM increment exhibit diurnal changes. However, the 30-minute plasma cortisol level remains unchanged throughout the day so that only this single criterion should be used (3).

Parenteral drug products should be inspected visually for particulate matter and discoloration whenever solution and container permit. Reconstituted CORTROSYNTM should not be retained.

#### **HOW SUPPLIED**

Box of 10 vials of CORTROSYN TM (cosyntropin) for Injection 0.25 mg NDC # 0548-5900-00

### Storage

Store at 15-30°C (59-86°F).

CORTROSYNTM is intended as a single dose injection and contains no antimicrobial preservative. Any unused portion should be discarded.

## Rx only

## **REFERENCES**

- 1. Wood, J.B. et al. LANCET 1.243, 1965.
- 2. Greig, W.R. et al. J. ENDOCR 34.411, 1966.
- 3. McGill, P.E. et al. ANN RHEUM DIS 26.123, 1967.

Amphastar Pharmaceuticals, Inc. Rancho Cucamonga, CA 91730 U.S.A. REV. 9-05

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

APPENDIX H: Investigator Brochure, Desoximetasone 0.15% Topical Spray

An Open Label, Safety Study to Assess the Potential for Adrenal Suppression Following Treatment with Desoximetasone 0.15% Topical Spray (Taro Pharmaceuticals U.S.A., Inc.) in Patients with Plaque Psoriasis

# **APPENDIX I: Protocol Revisions**

| Revisions | Revision Number | Revision Date |
|---|---|---|
| Protocol Rev Date added | 1 | 6/27/16 |
| to Title page, updated in footer and signature | | |
| page. | | |
| Blood draw volume | | |
| updated in Appendix C | | |
| <ul> <li>Clerical corrections</li> </ul> | | |
| made throughout the | | |
| document | | |

| Revisions | Revision Number | Revision Date |
|---|---|---|
| <ul> <li>Application Site Reactions were added to the protocol (Appendix C)</li> <li>Clerical corrections made throughout the document</li> <li>Protocol Revsion (Appendix I) updated</li> </ul> | 2 | 09/06/16 |